CLINICAL TRIAL: NCT05088772
Title: Pulmonary Function Following Hyperbaric Oxygen Therapy: A Prospective Cohort Study
Brief Title: Pulmonary Function After Hyperbaric Oxygen Therapy
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Connor Brenna, Resident Physician, University of Toronto
Other Study IDs: HBOT-PFT-19-5081.1
Record Dates: First submitted 2021-09-15; First posted 2021-10-22 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Oxygen Toxicity
Keywords: Hyperbaric Oxygen Therapy; Pulmonary Function; Hyperoxia
MeSH Terms: conditions — Hyperoxia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Hyperbaric Oxygen Therapy - Experimental Group: Patients receiving hyperbaric oxygen therapy at the Hyperbaric Medicine Unit (University Health Network, Toronto, ON, Canada)
  Interventions: Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy performed at 100% oxygen at 2.0-2.4 ATA, with 1-3 "air breaks", typically at 5 sessions per week, with limited variation depending on the treatment indication and patient/clinician preference.

SUMMARY:
Patients receiving hyperbaric oxygen therapy (HBOT) for any indication at the Hyperbaric Medicine Unit (University Health Network, Toronto, ON, Canada) from 2016-2021 were recruited to this prospective cohort study. While receiving HBOT (at 2.0-2.4 ATA, with 1-3 "air breaks", with specific treatment details determined on a case-by-case basis and directed by the clinical team), enrolled patients underwent pulmonary function testing prior to HBOT treatment and serially after each 20 completed treatment cycles.

DETAILED DESCRIPTION:
Patients receiving hyperbaric oxygen therapy (HBOT) at the Hyperbaric Medicine Unit (University Health Network, Toronto, ON, Canada) from 2016-2021 were recruited with informed consent to this prospective cohort study. All included patients underwent HBOT in one of three monoplace chambers (Sechrist 3600H and Sechrist 4100H, Sechrist Industries Inc., Anaheim, CA, USA; PAH-S1-3200, Pan-America Hyperbarics Inc., Plano, TX, USA) or via a plastic hood in a multiplace chamber (Hyperbaric System, Fink Engineering PTY-LTD, Warana, Australia). HBOT was performed with 100% oxygen at 2.0-2.4 ATA, with 1-3 "air breaks", typically at 5 sessions per week, with limited variation depending on the treatment indication and patient/clinician decision.

Study participants completed pulmonary function testing (PFTs) at several intervals during their HBOT treatment: prior to the first HBOT session, and serially after every 20 subsequent treatments. PFTs were performed using a KoKo Trek USB Spirometer software and pneumotachometer (KoKo, USA), with the assistance of a trained technician and in accordance with industry norms.

Retrospectively, PFT data was collected from all enrolled patients' electronic and paper medical charts. This data included anonymized patient demographics, as well as percentage of predicted forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and forced mid-expiratory flow rates (FEF25-75). PFT values underwent statistical analysis to identify potential effects of HBOT on pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to receive at least ten cycles of HBOT (for any indication)

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing HBOT at the investigators' large referral center, for any clinical indication.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD FRCPC, Principal Investigator — Hyperbaric Medicine Unit, University Health Network, Toronto, ON, Canada
Locations (1):
- Hyperbaric Medicine Unit, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brenna CTA, Khan S, Djaiani G, Au D, Schiavo S, Wahaj M, Janisse R, Katznelson R. Pulmonary function following hyperbaric oxygen therapy: A longitudinal observational study. PLoS One. 2023 May 31;18(5):e0285830. doi: 10.1371/journal.pone.0285830. eCollection 2023. PMID 37256885

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperbaric Oxygen Therapy - Experimental Group
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyperbaric Oxygen Therapy - Experimental Group
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m*m] | 27.1 (10.3)
Comorbidities [Number; unit: total comorbidities] | 123
Medications [Number; unit: total medications] | 115
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 23
  Former Smoker | 16
  Never Smoker | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage Predicted Forced Expiratory Volume in One Second (FEV1%)
Description: Change from baseline FEV1% defined as the highest value selected from at least three satisfactory pulmonary function tests at each timepoint
Time Frame: The outcome measure was evaluated at baseline (pre-HBOT) and after four weeks (20 treatments), eight weeks (40 treatments), and twelve weeks (60 treatments)
Measure: Mean (95% Confidence Interval); unit: Percentage of FEV1
Arm/Group | Hyperbaric Oxygen Therapy - Experimental Group
Number analyzed (Participants) | 86
Percentage of FEV1
  Pre-HBOT | 88.0 [83.3 to 92.7]
  20 Treatments | 85.9 [81.2 to 90.6]
  40 Treatments | 87.4 [82.4 to 92.3]
  60 Treatments | 84.6 [77.7 to 91.5]

2. Primary Outcome: Change in Percentage Predicted Forced Vital Capacity (FVC%)
Description: Change from baseline FVC% defined as the highest value selected from at least three satisfactory pulmonary function tests at each timepoint
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of FVC
Arm/Group | Hyperbaric Oxygen Therapy - Experimental Group
Number analyzed (Participants) | 86
Percentage of FVC
  Pre-HBOT | 88.8 [83.7 to 94.0]
  20 Treatments | 86.9 [81.8 to 92.1]
  40 Treatments | 89.2 [83.8 to 94.5]
  60 Treatments | 85.9 [79.1 to 92.6]

3. Primary Outcome: Change in Percentage Predicted Forced Mid-Expiratory Flow Rate (FEF25-75%)
Description: Change from baseline FEF25-75% defined as the highest value selected from at least three satisfactory pulmonary function tests at each timepoint
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage of FEF25-75
Arm/Group | Hyperbaric Oxygen Therapy - Experimental Group
Number analyzed (Participants) | 86
Percentage of FEF25-75
  Pre-HBOT | 66.9 [57.3 to 76.5]
  20 Treatments | 66.7 [57.1 to 76.3]
  40 Treatments | 66.2 [56.4 to 76.0]
  60 Treatments | 64.6 [53.1 to 76.2]

4. Secondary Outcome: Pulmonary Complications Following Hyperbaric Oxygen Therapy
Description: Any recorded pulmonary complications of HBOT, including but not limited to lung barotrauma, air embolism, and pneumothorax, identified through retrospective chart review
Time Frame: From date of recruitment until the date of first documented pulmonary complication or most recent follow-up, whichever came first, assessed up to a maximum of 5 years from study recruitment
Measure: Number; unit: Pulmonary Complications
Arm/Group | Hyperbaric Oxygen Therapy - Experimental Group
Number analyzed (Participants) | 86
Pulmonary Complications | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Hyperbaric Oxygen Therapy - Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 53/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperbaric Oxygen Therapy - Experimental Group (N=86)
Ear Barotrauma (Ear and labyrinth disorders) | 17
Seizure (Nervous system disorders) | 2
Ocular Changes (Eye disorders) | 16
Anxiety (Psychiatric disorders) | 18
Congestive Heart Failure (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT05088772/Prot_SAP_000.pdf